CLINICAL TRIAL: NCT01789775
Title: Phase 3 Efficacy and Safety Study of CD07805/47 Topical Gel in Subjects With Facial Erythema of Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.40174
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CD07805/47 gel Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Drug: CD07805/47 gel
- CD07805/47 gel (Experimental): Intervention: Drug: CD07805/47 gel
  Interventions: Drug: CD07805/47 gel Placebo

INTERVENTIONS:
Drug: Drug: CD07805/47 gel
  Arms: CD07805/47 gel Placebo
Drug: CD07805/47 gel Placebo
  Arms: CD07805/47 gel

SUMMARY:
Phase 3 efficacy and safety study of CD07805/47 topical gel in subjects with facial erythema associated with rosacea. The study hypothesis is that CD07805/47 gel, applied topically once daily is more efficacious than vehicle and provides an acceptable safety profile in the treatment of facial erythema associated with rosacea

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female who is at least 18 years of age or older.
2. A clinical diagnosis of facial rosacea.
3. A Clinician Erythema Assessment (CEA) score of greater than or equal to 3 at Screening and at Baseline/Day 1 (prior to the study drug application).
4. A Patient Self Assessment (PSA) score of greater than or equal to 3 at Screening and at Baseline/Day 1 (prior to the study drug application).

Key Exclusion Criteria:

1. More than 20 facial inflammatory lesions of rosacea
2. Particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
3. Current treatment with monoamine oxidase (MAO) inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, or alpha agonists.
4. Less than 3 months stable dose treatment with tricyclic anti depressants, cardiac glycosides, beta blockers or other antihypertensive agents.
5. Current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- France (2):
  - Galderma Investigational Site, Montpellier
  - Galderma Investigational Site, Nice
- Russia (4):
  - Galderma Investigational Site, Chelyabinsk
  - Galderma Investigational Site, Moscow
  - Galderma Investigational Site, Saint Petersburg
  - Galderma Investigational Site, Yekaterinburg
- Galderma Investigational Site, Eskilstuna, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- CD07805/47 Gel Placebo: Placebo
  Drug: CD07805/47 gel
- CD07805/47 Gel: Intervention: Drug: CD07805/47 gel
  CD07805/47 gel Placebo
Period: Overall Study
Arm/Group | CD07805/47 Gel Placebo | CD07805/47 Gel
Started | 55 | 57
Completed | 53 | 50
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD07805/47 Gel Placebo | CD07805/47 Gel | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.1) | 43.2 (10.8) | 44.0 (11.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 56 | 107
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  France | 6 | 8 | 14
  Russian Federation | 46 | 46 | 92
  Sweden | 3 | 3 | 6

OUTCOME MEASURES:

1. Secondary Outcome: Composite Success Assessment (CEA) and Patient Self Assessment(PSA).
Description: 30 Minutes Effect is defined as 1 grade improvement on CEA and PSA at 30 minutes.
Time Frame: D1
Reporting Status: Not Posted

2. Primary Outcome: Composite Success Assessment (CEA) and Patient Self Assessment(PSA).
Description: Composite Success is defined as 1-grade improvement on both Clinician Erythema Assessment (CEA) and Patient Self Assessment(PSA).
Time Frame: Day 29
Measure: Number; unit: participants
Arm/Group | CD07805/47 Gel Placebo | CD07805/47 Gel
Number analyzed (Participants) | 55 | 57
participants
  D29 Hour 3 | 32 | 48
  D29 Hour 5 | 33 | 46
  D29 Hour 7 | 35 | 43
  D29 Hour 9 | 33 | 39

ADVERSE EVENTS:
Arm/Group | CD07805/47 Gel Placebo | CD07805/47 Gel
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/57
Other Adverse Events (participants affected / at risk) | 0/55 | 10/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD07805/47 Gel Placebo (N=55) | CD07805/47 Gel (N=57)
Angiodema (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD07805/47 Gel Placebo (N=55) | CD07805/47 Gel (N=57)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No